CLINICAL TRIAL: NCT04934033
Title: Nice Healthy Brain - Cohort of Healthy People in Brain MRI, Together With a Language and Cognitive Assessment at the University Hospital of Nice
Brief Title: Cohort of Healthy People in Brain MRI, Together With a Language and Cognitive Assessment at the University Hospital of Nice
Acronym: NHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-AOI-01
Record Dates: First submitted 2021-06-09; First posted 2021-06-22 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Other): The participants will constitue a cohort of healthy volunteers, they will have a MRI, and language and cognitive assessment.
  Interventions: Other: Neurological assessments

INTERVENTIONS:
Other: Neurological assessments — The participants will have a MRI, and language and cognitive assessments.

SUMMARY:
The aim of this study is to constitute a cohort of healthy subjects in brain MRI, including functional and diffusion sequences, together with a language and cognitive assessment. This will make it possible to compare the data with those obtained in the same center and under the same examination conditions in brain tumor patients. The investigators seek to evidence general patterns of cerebral morphological and functional changes, correlated with behavioural scores, in brain-damaged patients.

ELIGIBILITY:
Inclusion Criteria:

* cerebral and psychiatric healthy volunteer
* agreeing to participate in this research
* 30 and 50 years old or between 60 and 75 years old

Exclusion Criteria:

* contra-indication to MRI
* refusal of patient participation
* pregnant, lactating or parturient women
* vulnerable people

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Number of cerebral MRI | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, Provence-Alpes-Côte d'Azur Region, France

IPD SHARING:
Plan to Share IPD: No